CLINICAL TRIAL: NCT03043001
Title: Using Memantine in Treating Bipolar Disorder Comorbid With Alcoholism
Brief Title: Memantine in Bipolar Patients With Alcoholism
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Ru-Band Lu, Distinguished Professor, National Cheng-Kung University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP_ALC_MM
Record Dates: First submitted 2017-01-26; First posted 2017-02-03 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: AOD Effects and Consequences
MeSH Terms: interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- add-on memantine therapy (Other): add-on memantine treatment
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — All the subjects will receive add-on memantine for 12 week
  Other Names: add-on therapy

SUMMARY:
Since memantine may not only inhibit overactivity of microglial cell, but also repair the damaged neurons and neurogenesis through activation of astroglial cell and release of neurotrophic factors, the investigators propose that the neurotrophic effect of memantine may benefit neurodegenerative diseases including bipolar disorders (BP) and alcohol dependence. In the current study, the investigator will investigate whether add-on memantine at a dose of 5 mg/day has a beneficial effect on BP comorbid with alcohol dependence.

DETAILED DESCRIPTION:
Each individual enter into this project will receive regulate treatment adding-on memantine medication. During each visit, patients will receive evaluation for their symptoms and plasma Brain-Derived Neurotropic Factor (BDNF), cytokines (e.g.., Interleukin-6(IL-6), IL-8) and neuropsychological performance.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient aged ≧18 and ≦65 years.
2. Signed informed consent by patient or legal representative.
3. The Chinese version of the modified Structural Interview of Affective Disorder and Schizophrenia-L(SADS-L), a semi-structured interview aimed at formulating the main bipolar II diagnoses based upon DSM-IV-TR criteria
4. A 2-day minimum for hypomania to diagnose BP.
5. Patient or a reliable caregiver was expected to ensure acceptable compliance and visit attendance for the duration of the study.

Exclusion Criteria:

1. Females who are pregnant or nursing.
2. Women of childbearing potential not using adequate contraception as per investigator judgment or not willing to comply with contraception for duration of study.
3. Patient has received memantine, other anti-inflammatory medication within 1 week prior to first dose of double-blind medication, such as cyclo-oxygenase 2 (Cox-2) inhibitors.
4. Clinically significant medical condition e.g., cardiac, hepatic and renal disease with current evidence of poor controlled.
5. Patient has received electroconvulsive therapy (ECT) within 4 weeks prior to the first dose of double-blind medication.
6. Increase in total SGOT, SGPT, BUN and creatinine by more than 3X upper limit of normal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
plasma BDNF change | baseline, week1, week2, week4, week8, week12
  treatment response change assessed by plasma BDNF

SECONDARY OUTCOMES:
attention change | baseline, 12-week
  attention change assessed by CPT
Side effect change | baseline, week1, week2, week4, week8, week12
  adverse effect change assessed by Side-Effects Checklist
cytokine level change | baseline, week1, week2, week4, week8, week12
  cytokine change assessed by cytokines level (IL-6, IL-8, IL-10)

OTHER OUTCOMES:
memory change | baseline, 12-week
  memory change assessed by WMS
executive function change | baseline, 12-week
  executive function change assessed by WCST

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Band Lu, MD, Principal Investigator — Department of Psychiatry, National Cheng Kung University
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No